CLINICAL TRIAL: NCT03461874
Title: Feasibility and Effectiveness of Acceptance and Commitment Therapy (ACT) for High Frequency Episodic Migraine Without Aura
Brief Title: ACT Therapy for HF Migraine
Acronym: ACTMigraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT protocol
Record Dates: First submitted 2018-02-15; First posted 2018-03-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Migraine Without Aura
Keywords: High-Frequency Migraine without aura; ACT
MeSH Terms: conditions — Migraine without Aura | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Education of patients followed by Pharmacological Prophylaxis, prescribed based on patients' profile (e.g. previous failures or contraindications), and limited to Topiramate, Propanolol, Amytriptiline or Calcium channel blockers
  Interventions: Behavioral: Education of patients; Drug: Pharmacological prophylaxis
- Treatment as usual + ACT (Experimental): Education of patients, Pharmacological Prophylaxis prescribed based on patients' profile, and eight group sessions of 90 minutes of ACT.
  The ACT consists in 6 weekly sessions, 90 minutes each, and 2 supplementary "booster" sessions, at two and four weeks after the conclusion of the weekly session. The main focus of the six ACT session will be the following: 1) Creative helplessness: the problem of control; 2) Indentifying values: introduction to Mindfulness; 3) Actions guided by values: working with thought; 4) Working with Acceptance and Willingness; 5) Committed Actions: self-as-context; 6) Integration: working with obstacles - wrap-up. The booster session starts with a mindfulness exercise, followed by a review of the contents covered across the ACT program.
  Interventions: Behavioral: Education of patients; Behavioral: ACT; Drug: Pharmacological prophylaxis

INTERVENTIONS:
Behavioral: Education of patients — During withdrawal treatment, patients are given recommendations on the approach to the use of drugs for acute treatment of migraine headache and on lifestyle issues. With regard to drugs, patients will be encouraged to restrict use of acute medications to headaches with "severe pain"; i.e., those rated as 8 or greater on a 0-10 (no pain - pain as bad as it could be). In these instances, patients will be instructed to take Eletriptan (40 mg) and/or Almotriptan (12.5 mg) as the first-line treatment, indomethacin (50 mg) as the second line, and will be specifically urged to avoid opioids. With regard to healthy lifestyle issues, patients will be encouraged to engage in moderate physical activity (i.e., 45 minutes twice per week of aerobic exercise), remain well hydrated, consume 3 meals per day, and maintain a regular sleep/wake pattern with at least 7-8 hours of sleep per night.
Behavioral: ACT — ACT consists in 6 weekly sessions, 90 minutes each, and 2 supplementary "booster" sessions, at two and four weeks after the conclusion of the weekly session. The main focus of the six ACT session will be the following: 1) Creative helplessness: the problem of control; 2) Indentifying values: introduction to Mindfulness; 3) Actions guided by values: working with thought; 4) Working with Acceptance and Willingness; 5) Committed Actions: self-as-context; 6) Integration: working with obstacles - wrap-up. The booster session starts with a mindfulness exercise, followed by a review of the contents covered across the ACT program.
  Patients will be trained in small groups (5-7 patients each) and guided by a specifically trained therapist. They will be educated to practice at home according to the instructions given by the therapist during the sessions.
  Arms: Treatment as usual + ACT
Drug: Pharmacological prophylaxis — Pharmacological prophylaxis will be prescribed based on patients' profile (e.g. previous failures or contraindications), and limited to Topiramate, Propanolol, Amytriptiline or Flunarizine. Doses will depend on patients' features, and the doses herein reported are to be intended as approximate ones: Topiramate at the dose of 50mg/day; Propanolol at the dose of 20mg/day; Amytriptiline at the dose of 10mg/day; Flunarizine at the dose of 5mg/day.

SUMMARY:
The aim is to compare the effectiveness of a behavioral treatment, the Acceptance and Commitment Therapy, provided as an add-on to the prophylactic treatment (treatment as usual-TaU) against TaU only on the reduction of monthly headaches frequency over 12 months in a sample of patients with high-frequency migraine without aura (i.e. reporting 9-14 days with headache per month in the previous three months).

ACT will be provided in small groups (5-7 patients each) by specifically trained therapists. The ACT consists in 6 weekly sessions, 90 minutes each, and 2 supplementary "booster" sessions, at two and four weeks after the conclusion of the weekly session. The main focus of the six ACT session will be the following: 1) Creative helplessness: the problem of control; 2) Identifying values: introduction to Mindfulness; 3) Actions guided by values: working with thought; 4) Working with Acceptance and Willingness; 5) Committed Actions: self-as-context; 6) Integration: working with obstacles - wrap-up. The booster session starts with a mindfulness exercise, followed by a review of the contents covered across the ACT program.

TaU will consist of education of patients, followed by pharmacological prophylaxis. Prophylaxis is prescribed based on patients' profile, such as previous failures, contraindications and so on by a neurologist with expertise in headache treatments and limited to Topiramate, Propanolol, Amytriptiline or Calcium channel blockers.

The study will be a Phase II Trial; randomized, Open-Label; Multicenter study. Patients will be randomized 1:1 to the two groups: 64 patients (32 per group) will be enrolled to detect an absolute difference of at least 2 migraine days/month in the experimental group (assuming alfa 5%, power 95%, up to 15% loss to follow-up).

DETAILED DESCRIPTION:
Background and significance. Patients with Migraine without Aura at high frequency of attacks (9/14 episode per month) are particularly exposed to the risk of medication overuse and chronification of their headache. The treatment of this category of patients can be difficult and they need a multidisciplinary treatment to learn techniques to manage their pain before than a chronic migraine condition has been induced. In recent years, non-pharmacological treatments have been proposed for treating patient with different forms of migraines and, among them, Mindfulness showed to be comparable to pharmacological prophylaxis.

ACT (Acceptance Commitment Therapy) belongs to the third wave of behavioral approaches used for different pathological conditions; the attention is focused on mental processes and the objective of this intervention is the psychological flexibility by cultivating six different positive psychological capacities; acceptance, defusion, sense of self, mindfulness, values, committed actions.

Reports in literature documented the effectiveness of ACT intervention to improve disability and impact in pain conditions and to develop the resilience of patients suffering from different physical or mental clinical problems. People with low resilience are exposed to have more emotional difficulties in terms of depression and anxiety and stress, in particular when they are suffering from chronic pain conditions such as migraine at high frequency, which has high impact on patients life. It has been demonstrated that specific interventions addressed to promote resilience can be helpful to reduce the impact of the disease and of pain. Studies on the use of mindfulness and ACT in particular in chronic pain conditions and migraine have demonstrated how these practices are helpful to tolerate pain, to contain the use of symptomatic medications and to modulate some specific characteristics of migraine patients personality, e.g. rigidity, low acceptance, low resilience.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. Diagnosis of High Frequency Episodic Migraine without Aura according to the IHS criteria, i.e. 9-14 days with headache per month in the previous three months.
3. Patients were stable in terms of pharmacological prophylaxis (for those cases in which it has been prescribed) in the preceding three months.

Exclusion Criteria:

1. Overuse of medications as defined by the ICHD, i.e. 15 or more NSAIDs per month, 10 or more triptans per month, 10 or more opioids, 10 or more combined compounds per month in the previous three months
2. Withdrawal intervention during the 18 months preceding the inclusion in the clinical program
3. Known major depression or other psychiatric condition as reported in clinical documentation
4. Known epilepsy and idiopathic intracranial hypertension as reported in clinical documentation
5. Psychotherapy (any approach) in the previous 18 months
6. Previous experience on mindfulness or meditation approaches (lifetime)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction of headaches frequency | 12 months
  Reduction of headaches frequency in patients treated by Pharmacological therapy only compared to patients treated by Pharmacological treatment + ACT

SECONDARY OUTCOMES:
Difference in the proportion of patients achieving the reduction of 50% or more of days with headache compared to baseline | 12 months
  Difference in the proportion of patients achieving the reduction of 50% or more of days with headache compared to baseline in the two groups.
Medications intake | 3, 6, 12 months
  Change in the number of medications for acute headaches treatment consumed.
Change in disability scores, assessed with the Migraine Disability Assessment. | 6, 12 months
  The Migraine Disability Assessment measures the impact of migraine headaches in terms of entirely missed workdays, partially missed workdays, entirely missed homework days, partially missed homework days and days with missed leisure/family activities. The score ranges between 0 and 270, with higher scores indicating higher disability; a score >=21 indicates presence of relevant disability.
Change in impact scores, assessed with the 6-item Headache Impact Test. | 6, 12 months
  The 6-item Headache Impact Test measures the impact of headaches on patients' ability to function on the job, at school, at home and in social situations. It is composed of six items, which are rated on a six-level scores (never, rarely, sometimes, very often, always, which are respectively assigned a score of 6, 8, 10, 11, 13). The total score is given by the sum of single items score and ranges between 36 and 78, with higher scores indicating worse impact. A total score below 46 indicates no impact; score in the range 50-55 indicates minor impact; score in the range 56-59 indicates substantial impact; score equal or higher than 60 indicate severe impact.
Change in in anxiety and depression scores, assessed with the Hospital Anxiety and Depression Scale. | 6, 12 months
  The Hospital Anxiety and Depression Scale has two separate score for depression and anxiety, each composed of seven items that are rated 0-3. Both anxiety and depression sub-scores are defined as the sum to the response to item and range between 0 and 21, with higher scores indicating worse anxiety and depression problems. A score >=8 is the cut-off for both anxiety and depression caseness.
Change in allodynia, assessed with the Allodynia Symptom Checklist. | 6, 12 months
  The Allodynia Symptom Checklist is composed of 12 items referring to the presence of allodynia, i.e. the clinical situation in which skin stimulation that ordinarily would not produce pain (e.g. wearing eyeglasses) is experienced as pain in the course of headache. Each item is rated on a 0-2 scale, and therefore the total checklist score is 0-24, with higher score indicating worse allodynia. Total score in the range 0-2 indicate no allodynia, those in the range 3-5 indicate mild allodynia, those in the range 6-8 indicate moderate allodynia and those >= 9 indicate severe allodynia.
Change in catastrophizing attitude, assessed with the Pain Catastrophizing Scale. | 6, 12 months
  The Pain Catastrophizing Scale is composed of 13 items, that have to be rated between 0 and 4. The total score is given by the sum of the response to the items and therefore ranges between 0 and 52, with higher scores indicating higher tendency to catastrophizing, and a score >= 30 indicates clinically relevant level of catastrophizing.
Change in acceptance attitude, assessed with the Acceptance & Action Questionnaire, second version. | 6, 12 months
  The Acceptance & Action Questionnaire-2 is composed of seven items addressing psychological inflexibility, each item ranges between 1 and 7, with higher scores indicating greater levels of inflexibility. The questionnaire score ranges between 7 and 49, and a score of 24 is a proposed cut-off.
Change in acceptance attitude, assessed with the Chronic Pain Acceptance Questionnaire. | 6, 12 months
  The Chronic Pain Acceptance Questionnaire is a measure of acceptance and experiential avoidance, defined in terms of the person's ability to participate daily activities while acknowledging the presence of pain, and to allow the experience of pain with no efforts to avoid or control it. It is composed of 20 items rated between 0 and 6, and the questionnaire total score is given by the sum to each of them. Score ranges between 0 and 120, with higher scores indicating higher capacity to engage in activities with presence of pain and with no attempts to avoid or control it.
Change in mindfulness, assessed with the Mindfulness Attention Awareness Scale. | 6, 12 months
  The scale measures people's tendency to be mindful of moment to moment experience, i.e. it focuses on the presence of attention and awareness of what occurs in the present. It is composed of 15 items, rated on a 1-6 scale: thus overall score ranges between 15 and 90, with higher scores reflecting higher mindfulness (i.e. higher attention and awareness of what occurs in the present).
Change in overall work productivity reduction. | 12 months
  Work productivity reduction is a composite measure given by two sub-dimension, namely absenteeism and presenteeism. Absenteeism is calculated as the number of days in which the person did not get to work because of headache. Presenteeism is calculated as the number of days in which the person was at work, but worked with reduced efficiency due to the presence of migraine headache. To calculate presenteeism, patients have to refer the number of days in which they worked with lower ability due to headache, and have to provide an estimate of their average performance level on a 1-99% scale. The portion needed to reach 100% performance is the productivity reduction coefficient, which is multiplied by the number of days with presenteeism to get the overall presenteeism measure.
  The overall work productivity reduction is given by the sum of absenteeism and presenteeism.
Risk of CM development | 12, 24 and 36 months
  Proportion of patients meeting the criteria for Chronic Migraine and Medication Overuse Headache (1.3 and 8.2 of the ICHD-3beta).

CONTACTS AND LOCATIONS:
Overall Officials: Licia Grazzi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrasik F, Grazzi L, D'Amico D, Sansone E, Leonardi M, Raggi A, Salgado-Garcia F. Mindfulness and headache: A "new" old treatment, with new findings. Cephalalgia. 2016 Oct;36(12):1192-1205. doi: 10.1177/0333102416667023. Epub 2016 Oct 1. PMID 27694139
- [Background] Giannini G, Zanigni S, Grimaldi D, Melotti R, Pierangeli G, Cortelli P, Cevoli S. Cephalalgiaphobia as a feature of high-frequency migraine: a pilot study. J Headache Pain. 2013 Jun 10;14(1):49. doi: 10.1186/1129-2377-14-49. PMID 23759110
- [Background] Grazzi L, Sansone E, Raggi A, D'Amico D, De Giorgio A, Leonardi M, De Torres L, Salgado-Garcia F, Andrasik F. Mindfulness and pharmacological prophylaxis after withdrawal from medication overuse in patients with Chronic Migraine: an effectiveness trial with a one-year follow-up. J Headache Pain. 2017 Dec;18(1):15. doi: 10.1186/s10194-017-0728-z. Epub 2017 Feb 4. PMID 28161874
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Luciano JV, Guallar JA, Aguado J, Lopez-Del-Hoyo Y, Olivan B, Magallon R, Alda M, Serrano-Blanco A, Gili M, Garcia-Campayo J. Effectiveness of group acceptance and commitment therapy for fibromyalgia: a 6-month randomized controlled trial (EFFIGACT study). Pain. 2014 Apr;155(4):693-702. doi: 10.1016/j.pain.2013.12.029. Epub 2013 Dec 28. PMID 24378880